CLINICAL TRIAL: NCT05436678
Title: An Open Label, Randomized, Multiple-Dose, Two-Treatment, Two-Period, Two-Sequence, Crossover Study to Evaluate the Comparative Bioavailability of PrimeC (Ciprofloxacin and Celecoxib) Tablets to Ciprofloxacin Tablets Co-administered With Celecoxib Capsules, in Healthy Adult Subject
Brief Title: A Multiple-Dose PK Study to Evaluate the Comparative Bioavailability of PrimeC Tablets to Ciprofloxacin Tablets Co-administered With Celecoxib Capsules, in Healthy Adult Subject
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: NeuroSense Therapeutics Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NST-PK-003
Record Dates: First submitted 2022-06-22; First posted 2022-06-29 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2022-06

CONDITIONS: Pharmacokinetics
MeSH Terms: interventions — Ciprofloxacin; Celecoxib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- PrimeC (Active Comparator): 2 PrimeC tablets (total single dose 748 mg) twice daily for 6.5 days following a meal
  Interventions: Drug: PrimeC 748 mg
- Marketed ciprofloxacin and celecoxib (Active Comparator): 750 mg of ciprofloxacin and 200 mg of celecoxib, co-administered twice daily for 6.5 days following a meal
  Interventions: Drug: Ciprofloxacin 750 MG; Drug: Celecoxib 200mg

INTERVENTIONS:
Drug: PrimeC 748 mg — PrimeC is an extended release formulation of a fixed dose combination of ciprofloxacin and celecoxib
  Arms: PrimeC
Drug: Ciprofloxacin 750 MG — Ciprofloxacin
  Arms: Marketed ciprofloxacin and celecoxib
Drug: Celecoxib 200mg — Celecoxib
  Arms: Marketed ciprofloxacin and celecoxib

SUMMARY:
This is an open-label, randomized, multiple-dose, two-treatment, two-period crossover study comparing the test and reference products. In each period of the study, either 2 × PrimeC tablets or reference products (ciprofloxacin co-administered celecoxib) will be administered to subjects every 12 hours for 6.5 days (13 total administrations), in fed conditions.

The subjects will receive the test treatment in one of the study periods and the reference treatment in the other study period according to a two-sequence randomization schedule. Blood samples will be collected before the morning dose on Day 1, before the morning and evening dose on Days 5 and 6, before the morning dose on Day 7 and at intervals over 48 hours after the morning dose on Day 7 (see Section 7.6) in each study period. Subjects will be confined at the clinical facility from at least 10.5 hours before the initial dose on Day 1 until approximately 48 hours after the final dose on Day 7.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, 18-55 years of age, inclusive, with a Body Mass Index (BMI) of 18.5-29.9 kg/m², inclusive.
2. Female subjects must meet at least one of the following criterion:

   * Agree to abstain from sexual intercourse from screening and throughout the duration of the study, with a documented secondary contraceptive method.
   * Have used and agree to continue to use a reliable method of contraception (e.g., hormonal contraceptives, condom with spermicide, IUD) for at least 30 days before initial dosing and throughout the duration of the study.
   * Surgically sterile (bilateral oophorectomy or hysterectomy, bilateral tubal ligation at least 3 months before initial dosing or Essure® device placement before the year 2018).
   * At least 1 year
3. Good health as determined by lack of clinically significant abnormalities in health assessments performed at screening.
4. Signed and dated informed consent form, which meets all criteria of current FDA regulations.
5. Subject understands the requirements of the study and is willing to comply with all study requirements.

Exclusion Criteria:

1. Females who are pregnant, lactating or likely to become pregnant during the study.
2. History of allergy or hypersensitivity to ciprofloxacin or other fluoroquinolones, celecoxib or other NSAIDs, any component of the study products, or history of any drug hypersensitivity or intolerance which, in the opinion of the Investigator, would compromise the safety of the subject or the study.
3. Significant history or current evidence of chronic infectious disease, system disorders, organ dysfunction especially cardiovascular disorders (e.g., heart failure, edema), respiratory disorders (e.g., asthma), hypertension, renal or hepatic disorders, diabetes or obesity.
4. QTc interval > 450 msec for males or > 470 msec for females or any clinically significant ECG abnormalities that, in the Investigator's opinion, would compromise the subject's safety for inclusion in the study. Significant history or current evidence of risk factors for Torsade de Pointes (TdP) (e.g., cardiac disease, heart failure, clinically significant hypokalemia or other electrolyte disorders, family history of Long QT Syndrome), as determined by the Investigator.
5. History or current evidence of myasthenia gravis or myasthenic syndrome.
6. History or current evidence of epilepsy, other seizures disorders, or other risk factors that may predispose to seizures or lower the seizure threshold; tendinitis or tendon rupture; peripheral neuropathy or aortic aneurysms.
7. Significant acute illness (e.g. acute infection) within 14 days before initial dosing, as determined by the Investigator.
8. Clinically significant history or presence of gastrointestinal disease (e.g., peptic ulcer, gastrointestinal bleeding) or history of malabsorption within the last year, as determined by the Investigator.
9. History of psychiatric disorders (e.g., anxiety, depression, insomnia, confusion) occurring within the last two years, which required the subject to be hospitalized or treated with medication.
10. Presence of a medical condition requiring regular treatment with prescription drugs (except hormonal contraceptives).
11. Use of pharmacologic agents (prescription or over-the-counter) or herbal products known or suspected to induce or inhibit drug-metabolizing enzymes (especially inducers and inhibitors of CYP1A2 and CYP2C9) within 30 days before initial dosing.
12. Use of dietary products (e.g., grapefruit products of all types) known or suspected to induce or inhibit drug-metabolizing enzymes (especially inducers and inhibitors of CYP1A2 and CYP2C9) within 14 days before initial dosing.
13. Use of any prescription medications (other than hormonal contraceptives and those noted above), especially prescription medications implicated in TdP or cardiac arrhythmia, terfenadine, pimozide, ergotamine; dihydroergotamine or over-the-counter medications implicated in TdP or cardiac arrhythmia; medications that interfere with hemostasis (e.g., warfarin, selective serotonin reuptake inhibitors, selective serotonin norepinephrine reuptake inhibitors), other quinolones, digoxin, and NSAIDs or antibiotics (all dosage forms and routes of administration; other than the study drugs) within 14 days before initial dosing.
14. Known or suspected to be a poor CYP2C9 metabolizer.
15. Receipt of any drug as part of a research study within 30 days before initial dosing or 5 half-lives, whichever is longer.
16. Drug or alcohol addiction, as determined by the Investigator, in the 12 months before initial dosing.
17. History of excessive alcohol consumption (on average more than 14 units of alcohol/week) during the past 12 months.
18. Donation or significant loss of whole blood (480 mL or more) within 30 days or plasma within 14 days before initial dosing.
19. Positive test results for HIV, Hepatitis B surface antigen, or Hepatitis C antibody.
20. Positive test results for drugs of abuse or cotinine at screening.
21. If female, has a positive pregnancy test at screening.
22. Use of tobacco- or nicotine-containing products within 90 days before initial dosing.
23. Difficulty swallowing capsules or tablets whole.
24. Unable or unwilling to comply with protocol restrictions and required study procedures.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
Cmax D1 | 1 day
  Maximum measured plasma concentration over the morning 12-hour dosing interval on Day 1.
Cmax D7 | 7 days
  Maximum measured plasma concentration over the morning 12-hour dosing interval on Day 7.
AUC0-12 D1 | 1 day
  Area under the plasma concentration versus time curve from time zero to the end of the morning 12-hour dosing interval on Day 1, as calculated by the linear trapezoidal method.
AUC0-12 D7 | 7 days
  Area under the plasma concentration time curve over the morning 12-hour dosing interval on Day 7, as calculated by the linear trapezoidal method.

SECONDARY OUTCOMES:
Cpre Dx | 7 days
  Measured pre-dose plasma concentration on Days 1, 5, 6 and 7; where D = Day 1, 5, 6 or 7; and x = m (morning dose) or e (evening dose).
Tmax D1 | 1 day
  Time of the maximum measured plasma concentration on Day 1 over the morning 12-hour dosing interval on Day 1.
AR Treatment R | 7 days
  For Treatment R (reference products), the ratio of accumulation over the morning 12-hour dosing interval on Day 7 compared the morning 12-hour dosing interval on Day 1 will be determined by the formula, (AUC0-12,D7 / AUC0-12,D1).
AR Treatment T | 7 days
  For Treatment T (PrimeC), the ratio of accumulation over the morning 12-hour dosing interval on Day 7 compared the morning 12-hour dosing interval on Day 1 will be determined by the formula, (AUC0-12,D7 / AUC0-12,D1).
Cav D7 | 7 days
  Average measured plasma concentration over the morning 12-hour dosing interval on Day 7.
Cmin D7 | 7 days
  Minimum measured plasma concentration over the morning 12-hour dosing interval on Day 7.
Ctrough D7 | 7 days
  Measured plasma concentration at the end of the morning dosing interval on Day 7.
Tmax D7 | 7 days
  Time of the maximum measured plasma concentration over the morning 12-hour dosing interval on Day 7.
λz | 7 days
  First order rate constant associated with the terminal (log-linear) portion of the curve following the last dose administered on the morning of Day 7.
t½ | 7 days
  The terminal half-life following the last dose administered on the morning of Day 7
Percent Fluctuation | 7 days
  Percent fluctuation over the morning 12-hour dosing interval on Day 7
Percent Swing | 7 days
  Percent swing over the morning 12-hour dosing interval on Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- Novum, Las Vegas, Nevada, United States